CLINICAL TRIAL: NCT04841408
Title: Prospective, Monocentric, Interventional Study on Spontaneous Vaginal Clearance of Mycoplasma Genitalium
Acronym: MYCOCLEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2021/06
Record Dates: First submitted 2021-04-07; First posted 2021-04-12 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Mycoplasma Genitalium Infection
Keywords: Mycoplasma genitalium; abortion; clearance; IST

STUDY DESIGN:
Intervention Model Description: Vaginal self-sampling performed by the patient at the follow-up visit at 3 weeks and remote follow-up at 9 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vaginal self-sampling (Experimental): Vaginal self-sampling performed by the patient at the follow-up visit at 3 weeks and remote follow-up at 9 weeks.
  Interventions: Other: Vaginal self-sampling

INTERVENTIONS:
Other: Vaginal self-sampling — Vaginal self-sampling performed by the patient at the follow-up visit at 3 weeks and remote follow-up at 9 weeks.

SUMMARY:
It is a prospective, monocentric, interventional study on spontaneous vaginal clearance of Mycoplasma genitalium.

The main objective is to evaluate the spontaneous vaginal clearance of M. genitalium in patients coming to perform a voluntary termination of pregnancy at the University Hospital of Bordeaux at 9 weeks after a vaginal sample positive for M. genitalium

DETAILED DESCRIPTION:
Mycoplasma genitalium is a bacterium that colonizes female genital tract and can be responsible for sexually transmitted infection . M. genitalium can cause cervicitis and more rarely high genital infections.

In the vast majority of cases, presence of M. genitalium is not accompanied by any symptoms and women do not develop disease. Natural history of M. genitalium infection is not well documented. Some studies have shown a natural clearance of infection in women. The published work mainly concerns patients at very high risk of sexually transmitted disease, but we do not have French data.

We propose to study the natural clearance of M. genitalium infection in patients consulting at the Orthogeny Centre of the University Hospital of Bordeaux. Results of this work will allow us to have a better knowledge of the natural history of M. genitalium infection.

ELIGIBILITY:
Inclusion Criteria:

* Patient selected during the first consultation, pre-abortion, and having a vaginal swab positive to M. genitalium.
* Patient hospitalized for an abortion at the University Hospital of Bordeaux.
* An affiliated patient or beneficiary of a social security system.
* Signing free and informed consent.

Exclusion criteria:

* Patient with vaginal co-infection with C. trachomatis.
* Patient with symptoms of high genital infection.
* Taking fluoroquinolones, macrolides or tetracyclines within 21 days of inclusion.
* Patient under legal protection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
clearance at week 3 | Week 3
  The clearance will be defined by a negative PCR test for M. genitalium in the vaginal sample taken at week 3.

SECONDARY OUTCOMES:
clearance at week 9 | Week 9
  The clearance defined by a negative PCR test for M. genitalium in the vaginal sample taken at week 9.
Prevalence of N. gonorrhoeae infections | Week 3, Week 9
  Prevalence of infections with N. gonorrhoeae calculated by making the ratio between the number of patients with a positive vaginal swab for N. gonorrhoeae compared to the total number of patients tested.
Prevalence of C. trachomatis infections | Week 3, Week 9
  Prevalence of infections with C. trachomatis calculated by making the ratio between the number of patients with a positive vaginal swab for C. trachomatis compared to the total number of patients tested.
Prevalence of M. genitalium infections | Week 3, Week 9
  Prevalence of infections with M. genitalium, calculated by making the ratio between the number of patients with a positive vaginal swab for M. genitalium compared to the total number of patients tested.
patient's sex life | Week 3, Week 9
  patient's sex life, assessed by a self-questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Bordeaux, Bordeaux, France

REFERENCES:
- [Derived] Berdoyes M, Bebear C, Roy CL, Balcon C, Hocke C, Baita D, Peuchant O. Spontaneous Clearance of Vaginal Mycoplasma genitalium in Women Undergoing Pregnancy Termination: A Prospective Cohort Study. BJOG. 2026 Jan 7. doi: 10.1111/1471-0528.70151. Online ahead of print. PMID 41502158